CLINICAL TRIAL: NCT04603352
Title: Impact of an Orthotic Garment on Gross Motor Skill Acquisition for Infants With Down Syndrome
Brief Title: Impact of an Orthotic Garment on Gross Motor Skills for Infants With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Principal Investigator, Megan Flores, Assistant Professor, University of St. Augustine for Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Down Syndrome Hip Helpers
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Gross motor function; home program; orthotic garment
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: This prospective, exploratory research study will employ a randomized controlled trial research design. The independent variables will be two conditions: usual care with the addition of a Hip Helpers® orthotic garment home program and usual care with no addition to the home program. The dependent variable will be an assessment of gross motor function over time as measured by the GMFM-88. Participants will be tested on the GMFM-88 each month, regardless of group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: Hip Helpers home program (Experimental): Participants in the intervention group will be given a custom pair of Hip Helpers® to use at home. Parents will begin the Hip Helpers® home program upon study entry and stop the program once the child is able to pull to stand independently. The Hip Helpers® home program protocol, which consists of using the orthotic garment twice daily for 30 minutes each time, will be given to the parents and supervised by the physical therapist. The Hip Helpers® should be donned when the child is actively playing, and not used sleep or when child is inactive.
  Interventions: Other: Hip Helpers home program
- Control group: No additional home program (No Intervention): Participants assigned to the control group will continue with their usual care.

INTERVENTIONS:
Other: Hip Helpers home program — Home program: Infants will wear Hip Helpers 30 minutes, twice per day.
  Other Names: Orthotic garment home program
  Arms: Intervention group: Hip Helpers home program

SUMMARY:
Infants with Down syndrome (DS) develop slower than their typically developing peers. Physical therapist (PT) supervised home programs have the potential to optimize gross motor development in a financially feasible way. An inexpensive orthotic garment (Hip Helpers®) is commonly employed by PTs as a home program supplement, but its effectiveness has not yet been investigated. The garment is worn as pliable shorts over a child's lower extremities to keep upper legs together, promoting a narrow base of support. This encourages activation of upright postural muscles to improve gross motor skill development. The purpose of this randomized controlled study is to investigate the impact of a home program using the Hip Helpers® orthotic garment on gross motor skill acquisition in infants with DS. We hypothesize that the addition of a structured home program using Hip Helpers®, supervised by a PT and implemented by parents, will increase the rate at which infants with DS acquire gross motor skills. Thirty-four participants, consisting of children who are at least three-months-old and are not yet able maintain sitting independently, will be randomly assigned to a control (n=17) or intervention group (n=17). PTs at pediatric therapy agencies will initiate the home program and administer the Gross Motor Function Measure-88 (GMFM-88) at regular intervals to monitor gross motor skill acquisition until the child is able to take three independent steps. Groups will be compared on the length of time elapsed between the acquisition of identified gross motor skills using independent t-tests. GMFM-88 scores will be compared between the two groups at different ages to identify trends using independent t-tests. The contribution of this project will be significant by informing physical therapists about the effectiveness of an inexpensive orthotic garment used in a supervised home program on gross motor outcomes in infants with DS.

DETAILED DESCRIPTION:
PTs at local Early Intervention and pediatric home health agencies will be recruited to administer the home program and GMFM-88 (Appendix D) tests on their patients that consent to participate in the study.

Recruitment of PTs will occur through an email sent to the local agencies. (Appendix E) The PTs (additional personnel) will watch a GMFM-88 training video. They will be given a GMFM-88 manual, and blank protocols.

Recruitment of participants will occur by the PTs, who are treating patients in a home health environment. The PTs will offer the opportunity to participate in the study to any of their patients/clients that meet the inclusion criteria by handing them a flyer about the study (Appendix A. If the parent of the potential participant is interested, the PT will ask the parent to call or email the closest investigator for more information (Austin, TX, San Marcos, CA, or St. Augustine, FL). The study investigator will discuss the study with the parent and, if parents decide to participate, email the informed consent to the parent. Parents who choose to participate will sign the informed consent form, which a study investigator will read and explain to the parents over the phone if requested. The parent will sign the informed consent in front of an investigator or the additional personnel PT.

PTs will take a course on the responsible conduct of research through CITI. They will also be trained by one of the investigators on the protocol of how to properly conduct the study. The investigator will instruct the PTs that they may not coerce or discuss the study with potential participants, but can only hand the recruitment flyer to the parent of the participant. The PT will not ask the parent about their participation further after handing them the flyer. If the parent has questions, the PT will instruct the parent to contact the investigator for more information. The PT will also be instructed that data collection will not begin until the parent has signed the informed consent and the investigator has given the participant a number and randomly assigned the participant to a group.

Parental consent will be obtained prior to any data collection. (Appendix C) Parents will complete a short demographic survey about their children (Appendix F).

The primary investigator (PI) will then assign the child a participant number and randomly assign the child to either the control group or the intervention group. This will be done using a randomization website: https://www.graphpad.com/quickcalcs/randomize1.cfm.

Once the child has been given a participant number and is assigned to a group, the PT will administer the first GMFM-88. PTs will continue to administer the GMFM-88 every 4 weeks to all participants, regardless of group. Each GMFM-88 testing session is expected to take approximately 20 minutes per session. PTs will stop administering the GMFM-88 when the child is able to take three independent steps. Additionally, PTs will note the child's age (in months/days) upon successfully attaining the following gross motor skills: 1) rolling, 2) sitting for 30 seconds independently, 3) transitioning from supine to sitting, 4) pulling up to stand, 5) standing independently for 30 seconds, 6) walking independently for three consecutive steps.

When a child gains one of these gross motor skills listed above, parents will be asked to obtain a short video of the child performing the skill using their smart phone or computer. Parents will email the video to the PI via an encrypted email. No additional data will be collected and transmitted with the video clips. The PI will instruct parents on how to send an encrypted email by going to this website for instructions: https://www.pandasecurity.com/mediacenter/panda-security/how-to-encrypt-email/. Data obtained by the PTs will be sent to the PI electronically using the participant's number only, with no other identifying information. The PI will label the videos sent by the parents with the participant's number and no other identifying information prior to saving them on a password-secured external hard drive. All de-identified data (including videos) will be stored on a password-secured external hard drive. Only the PI will have access to the hard drive. Signed consent/assent forms will be kept in a locked cabinet in the locked office of the PI for at least 3 years.

- Participants assigned to the control group will continue with their usual care.

Participants in the intervention group will be given a custom pair of Hip Helpers® to use at home. (Appendix G) Parents will begin the Hip Helpers® home program upon study entry and stop the program once the child is able to pull to stand independently. The Hip Helpers® home program protocol (Appendix H), which consists of using the orthotic garment twice daily for 30 minutes each time, will be given to the parents and supervised by the PT. The Hip Helpers® should be donned when the child is actively playing, and not used sleep or when child is inactive. To monitor compliance, parents will be given a log (Appendix I) which they will fill out and turn into the PT during each GMFM-88 assessment. The PT will give the log and the GMFM-88 scores with the participant's number to the PI each month. Additionally, PTs will supervise the home program, adjusting it as needed for their individual patients within the following parameters: 1) the target for total wear time should be 1 hour to be distributed throughout the day, 2) total wear time should not exceed 1 hour per day, 3) PT may suggest positions or activities to engage the child while wearing the garment, but may not suggest using while sleeping, 4) PT may "ramp up" wear time as needed for the individual participant starting with as little as 15 minutes per day and increasing to the full 1 hour per day.

Data collected by the PTs will be analyzed using IBM SPSS Statistics 24 software (IBM Corporation, Armonk, New York). To test the hypothesis that participants in the intervention group will improve their gross motor skills faster than participants in the control, groups will be compared on the length of time elapsed between the acquisition of identified gross motor skills using independent t-tests. A p-value < 0.05 will indicate significance. GMFM-88 scores will be compared between the two groups at different ages to identify trends using independent t-tests. Average percent improvement will be calculated for both groups on various domains of the GMFM-88, and the difference in these improvements will be calculated between the two groups.

Videos will be qualitatively analyzed by coding and triangulation. Quality and variability of movement will be coded by 2 of the investigators for each video. Inter- and intrarater agreement will be established before formal data coding using a ratio of agreements/ disagreements x 100 to establish a percentage of agreements. Short descriptions of movement quality will be written by 2 investigators with all 3 investigators coding and categorizing the descriptions to determine emergent themes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of DS
* between the ages of three to nine months
* not able to maintain upright sitting independently

Exclusion Criteria:

* a diagnosis unrelated to DS that limits gross motor movement
* medical restrictions that contraindicate movement
* a history of hip displacement or dislocation

Ages: 3 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure - 88 (GMFM-88 | Assessed every 4 weeks from randomization until child takes three independent steps, up to 36 months
  The GMFM-88 is a measure of gross motor function for children with Down syndrome (DS) under six years old. The examiner scores a child's capabilities across five dimensions of functional movement: A) Lying and Rolling, B) Sitting, C) Crawling and Kneeling, D) Standing, and E) Walking, Running, and Jumping. Each dimension consists of several items on an ordinal scale. The child receives a score of 0 (does not initiate), 1 (initiates), 2 (partially completes), or 3 (completes). This outcome measure can be administered by direct observation or by parent report. For children with DS, the GMFM-88 has strong interrater reliability (ICC = 0.9

SECONDARY OUTCOMES:
Incidence of gross motor milestone achievement, by parent report | From date of randomization at each documented progression until child takes three independent steps, assessed up to 36 months.
  Short videos will be taken by parents at achievement of gross motor milestones.

CONTACTS AND LOCATIONS:
Overall Officials: Megan B Flores, PT, MPT, PhD, Principal Investigator — University of St. Augustine for Health Sciences
Locations (3):
- United States (3):
  - University of St. Augustine for Health Sciences, San Marcos, California
  - University of St. Augustine for Health Sciences, Saint Augustine, Florida
  - University of St. Augustine for Health Sciences, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palisano RJ, Walter SD, Russell DJ, Rosenbaum PL, Gemus M, Galuppi BE, Cunningham L. Gross motor function of children with down syndrome: creation of motor growth curves. Arch Phys Med Rehabil. 2001 Apr;82(4):494-500. doi: 10.1053/apmr.2001.21956. PMID 11295010
- [Background] Pereira K, Basso RP, Lindquist AR, da Silva LG, Tudella E. Infants with Down syndrome: percentage and age for acquisition of gross motor skills. Res Dev Disabil. 2013 Mar;34(3):894-901. doi: 10.1016/j.ridd.2012.11.021. Epub 2013 Jan 2. PMID 23291506
- [Background] Tudella E, Pereira K, Basso RP, Savelsbergh GJ. Description of the motor development of 3-12 month old infants with Down syndrome: the influence of the postural body position. Res Dev Disabil. 2011 Sep-Oct;32(5):1514-20. doi: 10.1016/j.ridd.2011.01.046. Epub 2011 Mar 1. PMID 21367575
- [Background] Ulrich BD. Opportunities for early intervention based on theory, basic neuroscience, and clinical science. Phys Ther. 2010 Dec;90(12):1868-80. doi: 10.2522/ptj.20100040. Epub 2010 Oct 21. PMID 20966210
- [Background] Parker SE, Mai CT, Canfield MA, Rickard R, Wang Y, Meyer RE, Anderson P, Mason CA, Collins JS, Kirby RS, Correa A; National Birth Defects Prevention Network. Updated National Birth Prevalence estimates for selected birth defects in the United States, 2004-2006. Birth Defects Res A Clin Mol Teratol. 2010 Dec;88(12):1008-16. doi: 10.1002/bdra.20735. Epub 2010 Sep 28. PMID 20878909
- [Background] Knychala NAG, de Oliveira EA, de Araujo LB, de Oliviera Azevedo V. Influence of the home environment on the motor development of infants with Down syndrome. Fisioter Pesqui. 2018;25(2):202-208
- [Background] Houwen S, Visser L, van der Putten A, Vlaskamp C. The interrelationships between motor, cognitive, and language development in children with and without intellectual and developmental disabilities. Res Dev Disabil. 2016 Jun-Jul;53-54:19-31. doi: 10.1016/j.ridd.2016.01.012. Epub 2016 Feb 4. PMID 26851384
- [Background] Ulrich DA, Lloyd MC, Tiernan CW, Looper JE, Angulo-Barroso RM. Effects of intensity of treadmill training on developmental outcomes and stepping in infants with Down syndrome: a randomized trial. Phys Ther. 2008 Jan;88(1):114-22. doi: 10.2522/ptj.20070139. Epub 2007 Oct 16. PMID 17940103
- [Background] Wu J, Looper J, Ulrich BD, Ulrich DA, Angulo-Barroso RM. Exploring effects of different treadmill interventions on walking onset and gait patterns in infants with Down syndrome. Dev Med Child Neurol. 2007 Nov;49(11):839-45. doi: 10.1111/j.1469-8749.2007.00839.x. PMID 17979862
- [Background] Angulo-Barroso RM, Wu J, Ulrich DA. Long-term effect of different treadmill interventions on gait development in new walkers with Down syndrome. Gait Posture. 2008 Feb;27(2):231-8. doi: 10.1016/j.gaitpost.2007.03.014. Epub 2007 May 17. PMID 17499993
- [Background] Russell D, Palisano R, Walter S, Rosenbaum P, Gemus M, Gowland C, Galuppi B, Lane M. Evaluating motor function in children with Down syndrome: validity of the GMFM. Dev Med Child Neurol. 1998 Oct;40(10):693-701. doi: 10.1111/j.1469-8749.1998.tb12330.x. PMID 9851239
- [Background] Gemus M, Palisano R, Russell D, Rosenbaum P, Walter SD, Galuppi B, Lane M. Using the gross motor function measure to evaluate motor development in children with Down syndrome. Phys Occup Ther Pediatr. 2001;21(2-3):69-79. PMID 12029855
- [Background] Russell DJ, Rosenbaum PL, Cadman DT, Gowland C, Hardy S, Jarvis S. The gross motor function measure: a means to evaluate the effects of physical therapy. Dev Med Child Neurol. 1989 Jun;31(3):341-52. doi: 10.1111/j.1469-8749.1989.tb04003.x. PMID 2753238
- [Background] Silva LM, Schalock M, Garberg J, Smith CL. Qigong massage for motor skills in young children with cerebral palsy and Down syndrome. Am J Occup Ther. 2012 May-Jun;66(3):348-55. doi: 10.5014/ajot.2012.003541. PMID 22549600
- [Background] Palisano RJ, Kolobe TH, Haley SM, Lowes LP, Jones SL. Validity of the Peabody Developmental Gross Motor Scale as an evaluative measure of infants receiving physical therapy. Phys Ther. 1995 Nov;75(11):939-48; discussion 948-51. doi: 10.1093/ptj/75.11.939. PMID 7480124
- [Background] Ulrich DA, Ulrich BD, Angulo-Kinzler RM, Yun J. Treadmill training of infants with Down syndrome: evidence-based developmental outcomes. Pediatrics. 2001 Nov;108(5):E84. doi: 10.1542/peds.108.5.e84. PMID 11694668
- [Background] Capio CM, Mak TCT, Tse MA, Masters RSW. Fundamental movement skills and balance of children with Down syndrome. J Intellect Disabil Res. 2018 Mar;62(3):225-236. doi: 10.1111/jir.12458. Epub 2017 Dec 5. PMID 29205624
- [Background] Pin TW, Butler PB, Cheung HM, Shum SL. Relationship between segmental trunk control and gross motor development in typically developing infants aged from 4 to 12 months: a pilot study. BMC Pediatr. 2019 Nov 11;19(1):425. doi: 10.1186/s12887-019-1791-1. PMID 31711441
- [Background] Shumway-Cook A, Woollacott MH. Dynamics of postural control in the child with Down syndrome. Phys Ther. 1985 Sep;65(9):1315-22. doi: 10.1093/ptj/65.9.1315. PMID 3162178
- [Background] Wang HY, Long IM, Liu MF. Relationships between task-oriented postural control and motor ability in children and adolescents with Down syndrome. Res Dev Disabil. 2012 Nov-Dec;33(6):1792-8. doi: 10.1016/j.ridd.2012.05.002. Epub 2012 Jun 13. PMID 22699252
- [Background] de Graaf G, Buckley F, Skotko BG. Estimates of the live births, natural losses, and elective terminations with Down syndrome in the United States. Am J Med Genet A. 2015 Apr;167A(4):756-67. doi: 10.1002/ajmg.a.37001. PMID 25822844
- [Background] Boulet SL, Molinari NA, Grosse SD, Honein MA, Correa-Villasenor A. Health care expenditures for infants and young children with Down syndrome in a privately insured population. J Pediatr. 2008 Aug;153(2):241-6. doi: 10.1016/j.jpeds.2008.02.046. Epub 2008 Apr 23. PMID 18534234